CLINICAL TRIAL: NCT04279470
Title: Chimeric Antigen Receptor T-cell and Cellular Therapies for the Treatment of cAncer or BLood Diseases: Evaluation of Reporting of Adverse Events
Acronym: CARTABLE
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Principal Investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-20-01
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Adverse Drug Reactions; Cancer
Keywords: CAR-T cell; Cellular Therapies
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adverse Events with cellular therapies: Cases reported in the World Health Organization (WHO) and the French pharmacovigilance database of patients treated by Chimeric Antigen Receptor T-cell and Cellular Therapies, with a chronology compatible with the drug toxicity
  Interventions: Drug: CAR T-cell and Cellular Therapies

INTERVENTIONS:
Drug: CAR T-cell and Cellular Therapies — Chimeric Antigen Receptor T-cell and Cellular Therapies for the treatment of a cancer either solid or hematologic malignancy

SUMMARY:
CAR-T cells and cellular therapies may lead to various adverse reactions. This study investigates reports of different toxicities for cellular therapies in the World Health Organization's (WHO) global database of individual safety case reports (VigiBase).

DETAILED DESCRIPTION:
CAR-T cells and cellular therapies are responsible of a wide range of side effects.The investigators use VigiBase, the World Health Organization (WHO) database of individual safety case reports, to identify cases of adverse drug reactions following treatment with cellular therapies

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2020
* Adverse events reported were including any MedDRA terms
* Patients treated with cellular therapies reported in the WHO database.

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with cellular therapy for solid or hematologic cancer
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events with significant over-reporting CAR-T cells and other cellular therapies | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020
  Identification and report of various toxicities of cellular therapies.

SECONDARY OUTCOMES:
Causality assessment of reported adverse events according to the WHO system | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020
Description of the type of adverse event depending on the class and the target of cellular therapy | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020
Description of the duration of treatment when the toxicity happens and the time to onset | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020
Description of the population of patients having an adverse event | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dolladille C, Ederhy S, Ezine E, Choquet S, Nguyen LS, Alexandre J, Moslehi JJ, Dechartres A, Salem JE. Chimeric antigen receptor T-cells safety: A pharmacovigilance and meta-analysis study. Am J Hematol. 2021 Sep 1;96(9):1101-1111. doi: 10.1002/ajh.26259. Epub 2021 Jun 23. PMID 34057232